CLINICAL TRIAL: NCT03377855
Title: Addressing Origins of the Opioid Epidemic by Improving Prescribing for Opioid-Naive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York State Health Foundation (Unknown); The Institute for Family Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1710018646; 17-05047 (Other Grant/Funding Number: NYS Health Foundation)
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Opioid Use; Opioid-Related Disorders; Opioid Abuse; Prescription Drug Abuse and Dependency
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a interrupted time series study model with one study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Default Prescribing Change (Experimental): In the e-prescribing system, the default opioid dosage/duration is changed to the minimum recommended dosage from the CDC guidelines for short acting opioids.
  Interventions: Other: Default Prescribing Change

INTERVENTIONS:
Other: Default Prescribing Change — In the e-prescribing system, the default opioid dosage/duration is changed to the minimum recommended dosage from the CDC guidelines for short acting opioids.

SUMMARY:
Risk of long-term opioid dependence increases with initial opioid dose/duration, but despite recent Centers for Disease Control and Prevention (CDC)-endorsed minimum doses for initial opioid prescription, primary care providers are likely to overprescribe. In this quality improvement project, primary care departments at Weill Cornell and the Institute for Family Health (federally qualified health center in New York City) will implement an unobtrusive "nudge" in their electronic prescribing software to promote the CDC-endorsed low doses for all opioids. In the evaluation, we will employ a quasi-experimental design with rigorous interrupted time series analysis methods to assess the effect of the "nudge" on prescribing rates. The analysis will be performed at the provider level, with deidentified physician data and a limited data set (fully deidentified except for date of prescription) of patient-level data.

DETAILED DESCRIPTION:
The two participating institutions, WCMC (Weill Cornell Medical College) and IFH (Institute for Family Health), intend to redesign the e-prescribing interface to create a minor "nudge" to encourage prescribers to prescribe the minimum dose set by the 2016 CDC guideline for opioid-naive patients in 2018. The change to the e-prescribing system is that after a prescriber chooses the drug they wish to prescribe, the minimum recommended dosage from the CDC guidelines will be displayed. The prescriber can choose to change the dosage by overwriting in the field box. The changes to the prescriber system will be implemented at two Weill Cornell clinical organizations: Weill Cornell Internal Medicine Associates (WCIMA) and Weill Cornell Medical Associates (CMA), and at all locations at our collaborating institution IFH (Institute for Family Health). Weill Cornell and IFH will provide data for the analysis, which will be conducted by the co-investigators on this protocol. The project will assess data pre- and post- implementation to study prescribing patterns.

ELIGIBILITY:
Inclusion Criteria:

* Prescriber - practices internal medicine at WCMC OR family practice at IFH and has prescribed opioids since 11/1/2015

Exclusion Criteria:

* Prescriber - has not written any opioid prescriptions during the study period

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 948 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of opioid prescriptions for opioid-naïve patients that comply with CDC recommendations before and after the intervention | Two years prior to and six months after implementation
  Change in the proportion of opioid prescriptions for opioid-naïve patients that comply with CDC recommendations before and after the intervention

SECONDARY OUTCOMES:
Change in the average days of supply of opioids for opioid naive patients | Two years prior to and six months after implementation
  Change in the average days of supply of opioids for opioid naive patients

CONTACTS AND LOCATIONS:
Overall Officials: Jessica S Ancker, PhD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - The Institute for Family Health, New York, New York
  - Weill Medical College of Cornell University, New York, New York

IPD SHARING:
Plan to Share IPD: No
This data is protected by HIPAA and IRB/human subjects protections. In addition, the data is scheduled to be destroyed after publication of results.

REFERENCES:
- [Background] Malhotra S, Cheriff AD, Gossey JT, Cole CL, Kaushal R, Ancker JS. Effects of an e-Prescribing interface redesign on rates of generic drug prescribing: exploiting default options. J Am Med Inform Assoc. 2016 Sep;23(5):891-8. doi: 10.1093/jamia/ocv192. Epub 2016 Feb 17. PMID 26911828